CLINICAL TRIAL: NCT05348200
Title: A Randomized, Dose-Ranging, Double Blind Study to Demonstrate the Safety and Efficacy of a CITI-002 Cream in the Seven Day Twice-Daily Treatment of Grade II or III Hemorrhoids
Brief Title: Safety and Efficacy of CITI-002 in Adult Patients With Moderate Grade Hemorrhoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Citius Pharmaceuticals, Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 143-11351-202
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-04

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Lidocaine; halobetasol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in one of the 5 Treatment Groups in a 1:1:1:1:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Monad 1 cream (Active Comparator): Topical cream applied to the peri-anal area twice daily for seven days.
  Interventions: Drug: Monad 1
- Monad 2 cream (Active Comparator): Topical cream applied to the peri-anal area twice daily for seven days.
  Interventions: Drug: Monad 2
- Monad 3 cream (Active Comparator): Topical cream applied to the peri-anal area twice daily for seven days.
  Interventions: Drug: Monad 3
- Combination-CITI-002 (low dose) cream (Experimental): Topical cream applied to the peri-anal area twice daily for seven days.
  Interventions: Drug: Combination - CITI-002 (low dose)
- Combination-CITI-002 (high dose) cream (Experimental): Topical cream applied to the peri-anal area twice daily for seven days.
  Interventions: Drug: Combination - CITI-002 (high dose)

INTERVENTIONS:
Drug: Monad 1 — Single therapy cream containing Lidocaine. Lidocaine is a topical anesthetic.
  Other Names: Lidocaine
  Arms: Monad 1 cream
Drug: Monad 2 — Single therapy cream containing Halobetasol Propionate (low-strength). HPB is a topical corticosteroid.
  Other Names: Halobetasol Propionate (HBP)
  Arms: Monad 2 cream
Drug: Monad 3 — Single therapy cream containing Halobetasol Propionate (high strength).
  Other Names: Halobetasol Propionate
  Arms: Monad 3 cream
Drug: Combination - CITI-002 (low dose) — Combination cream containing Lidocaine and HBP (low)
  Other Names: CITI-002 L
  Arms: Combination-CITI-002 (low dose) cream
Drug: Combination - CITI-002 (high dose) — Combination cream containing Lidocaine and HBP (high)
  Other Names: CITI-002 H
  Arms: Combination-CITI-002 (high dose) cream

SUMMARY:
A Randomized Phase 2 double blind study which aims to determine the safety and efficacy of CITI-002 cream in adult patients with Goligher's grade II or III hemorrhoids.

DETAILED DESCRIPTION:
This Phase 2 study aims to compare the safety and efficacy of 5 different treatment groups. The study drug will be applied twice daily for 7 days. Response to the study drug will be measured through patient responses to an electronic Patient Reported Outcome (ePRO). There are 4 study visits: first visit is screening (day 1), follow-up visit (day 5), end of treatment (day 8), and end of study visit (day 15). There will also be one telephone visit on day 2. This study will be done in ~16 US sites and about 300 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female 18 years of age or older.
* Signs written informed consent for the study.
* Females must be post-menopausal , surgically sterile , or use an effective method of birth control, or women of childbearing potential (WOCBP) must have a negative Urine Pregnancy Test (UPT).
* Clinical diagnosis of confirmed symptomatic Goligher's classification Grade II or III hemorrhoids that are treatable without surgical intervention.
* Has an active "flare up" of hemorrhoids .
* Willing and able to apply the test article as directed, comply with study instructions, read, understand, and complete required questionnaires in English, and commit to all follow-up visits for the duration of the study.
* In good general health and free of any disease state or physical condition that might impair evaluation of hemorrhoids or exposes the subject to an unacceptable risk by study participation.
* If using stool softeners and/or fiber supplementation, must be on a stable regimen for at least 4 days prior to enrolling in the study and agree to remain on the stable regimen while in the study.
* Free of Coronavirus Disease (COVID) related signs and symptoms and if unvaccinated has no known close exposure to any person with COVID 10 days prior to enrolling in the study.
* Has access to device capable of communicating and interacting with daily data collection application (e.g., a smart phone capable of running the data collection application)

Exclusion Criteria:

* Has Grade I hemorrhoids; Grade III hemorrhoids that require surgical intervention; or Grade IV hemorrhoids.
* Females who are pregnant, lactating, or is planning to become pregnant during the study.
* Has anorectal condition(s) such as malignant tumors of the anus or rectum, fistula-in-ano or chronic sepsis, fissure(s), incontinence, or condylomata.
* Has a history of previous proctological surgery or has active inflammatory bowel disease.
* Used the following systemic, oral, or topical therapies for the periods specified prior to enrolling into the study:

  1. Within 1 day: topical application of any kind to the rectal/peri-anal area.
  2. Within 4 days: prescription (including topical steroids), over-the-counter (OTC), homeopathic, or home remedy treatments, including but not limited to, oral formulations, cream, ointment, gel, foam, sitz baths, wipes, or liquids labeled or intended for the treatment of hemorrhoids that could have a significant effect on the disease in the opinion of the investigator.
* If currently using aspirin (excluding low-dose for prophylaxis), has an uncorrected coagulation defect, or concurrently uses anticoagulants (except non-steroidals).
* Used systemic corticosteroids or narcotics within 4 weeks prior to Visit 1/Baseline.
* Currently enrolled in an investigational drug, biologic, or device study.
* Has used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to first application of the test article.
* History of sensitivity to any of the ingredients in the test articles.
* Has Addison's Disease, Cushing's Syndrome, or impaired Hypothalamic-Pituitary-Adrenal (HPA) axis function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Hemorrhoid symptoms | Day 8
  Change in hemorrhoidal symptoms (pain, burning, itching, and swelling) as measured by the patient using a numeric rating scale.

SECONDARY OUTCOMES:
Change in Hemorrhoidal bother. | Day 8
  Change of hemorrhoidal symptoms related to bowel movement interference and pressure as measured by the patient using a numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lader, PhD, Principal Investigator — Citius Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Site #01, Huntsville, Alabama
  - Site #07, Tucson, Arizona
  - Site #06, Chula Vista, California
  - Site #09, Pomona, California
  - Site #16, San Diego, California
  - Site #03, San Diego, California
  - Site #05, West Palm Beach, Florida
  - Site #10, Covington, Louisiana
  - Site #12, Prairieville, Louisiana
  - Site #02, Wyoming, Michigan
  - Site #14, Gulfport, Mississippi
  - Site #08, Omaha, Nebraska
  - Site #11, Mentor, Ohio
  - Site #13, Tulsa, Oklahoma
  - Site #04, Harrisburg, Pennsylvania
  - Site #15, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No